CLINICAL TRIAL: NCT07043608
Title: A Phase II Study of Zanzalintinib for Metastatic Clear Cell Renal Cell Carcinoma With Bone Metastases in Patients Previously Treated With Immune Checkpoint Inhibitors
Brief Title: Zanzalintinib for Metastatic Clear Cell Renal Cell Carcinoma With Bone Metastases
Acronym: ZAMBONI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kelly Fitzgerald, MD (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor-Investigator, Kelly Fitzgerald, MD, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25521; NCI-2025-04328 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Clear Cell Renal Cell Cancer (ccRCC); Clear Cell Renal Carcinoma; Clear Cell Renal Cell Carcinoma Metastatic; Clear Cell Renal Cancer; Bone Metastases of a Malignant Tumor; Clear Cell Renal Cell Carcinoma; Bone, Metastatic Cancer; Metastatic Cancer; Metastatic Renal Cell Carcinoma; Metastases to Bone
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma; Neoplasm Metastasis | interventions — Diphosphonates; Zoledronic Acid; Ibandronic Acid; Denosumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Zanzalintinib) (Experimental): Participants will receive 100 mg Zanzalintinib administered orally once a day in 28-day cycles, starting on cycle 1, day 1, and continued until criteria for removal from study are met. Investigator-choice bone-strengthening agent (BSA) will be selected and administered at a standard dose/interval starting within 30 days of cycle 1, day 1. Non-investigational RT for symptomatic metastases, including bone metastases, is allowed per investigator discretion. Participants must receive at least 1 dose of zanzalintinib prior to treatment pause for RT. Participants may continue study treatment until they are unable to tolerate treatment due to toxicity or demonstrate progression (per RECIST) from the time of initiating treatment.
  Interventions: Drug: Zanzalintinib; Drug: Investigator Choice of Bone Strengthening Agents (BSA); Radiation: Non-Investigational Radiation Therapy (RT); Procedure: Bone Scan; Procedure: Computerized tomography (CT) Scan

INTERVENTIONS:
Drug: Zanzalintinib — Given orally (PO)
  Other Names: XL092
Drug: Investigator Choice of Bone Strengthening Agents (BSA) — One BSA will be chosen, at the discretion of the investigator and given intravenously (IV)
  Other Names: Bisphosphonate; Receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitor; Zoledronic acid; Ibandronate; Denosumab
Radiation: Non-Investigational Radiation Therapy (RT) — Non-investigational RT is permitted for symptomatic bone metastases.
  Other Names: Standard-of-Care Radiation Therapy; Radiation Therapy; Non-Investigational RT
Procedure: Bone Scan — Undergo Bone Scan
Procedure: Computerized tomography (CT) Scan — Undergo Imaging

SUMMARY:
This is a single-institution, phase 2 trial of zanzalintinib plus investigator-choice bone-strengthening agent in patients with metastatic renal cell carcinoma (RCC) with bone metastases whose disease has advanced on 1-3 prior lines of therapy, including at least one immune oncology-based (IO) therapy in the adjuvant or first-line metastatic setting.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate progression-free survival (PFS) at 12 months in participants with RECIST-measurable metastatic RCC and bone metastases at baseline, and who have been previously treated with contemporary IO-based therapy.

SECONDARY OBJECTIVES:

I. To determine the rate of skeletal-related events (SRE).

II. To determine the rate of osteonecrosis of the jaw (ONJ).

III. To determine the rate of systemic toxicity.

IV. To determine median overall PFS.

V. To determine median overall survival (OS) in participants.

VI. To evaluate the objective response rate (ORR) in participants with measurable disease at baseline according to RECIST v 1.1.

VII. To evaluate PFS at 24 months in patients with Response Evaluation Criteria in Solid Tumors (RECIST)-measurable disease (metastatic RCC and bone metastases) at baseline.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of treatment on osseous microenvironment including immune and metabolic microenvironment using Flow cytometry, bulk Ribonucleic acid sequencing (RNA-seq), Single-cell RNA sequencing (scRNA-seq), Immunohistochemistry (IHC), spatial genomic and/or proteomic profiling.

II. Describe changes in quality of life (HRQoL) using European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30).

OUTLINE:

Participants will receive zanzalintinib and continue until criteria for removal from study are met. Investigator-choice bone-strengthening agent (BSA) will be administered at a standard dose/interval starting within 30 days of first study treatment. Non-investigational Radiation therapy (RT) for symptomatic metastases, including bone metastases, is allowed per investigator discretion. Participants may continue study treatment until unacceptable toxicity or demonstrated disease progression, or death whichever occurs first and followed for survival for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have unresectable advanced or metastatic RCC with a predominant clear cell histologic component .
2. At least three bone metastases are present and detectable on bone scan, and at least one bone metastasis is NOT planned to be treated with radiation therapy.
3. Previously treated with 1-3 prior lines of therapy in at least one of the following settings:

   1. Metastatic setting; must have received combination therapy containing either programmed cell death protein 1 (PD-1) inhibitor/cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor or PD-1 inhibitor/vascular endothelial growth factor receptor (VEGFR)-targeting tyrosine kinase inhibitors (TKI).
   2. Adjuvant setting; must have received pembrolizumab and have had documented progression of disease within 1 year of the first dose of pembrolizumab .
4. Age ≥18 years.
5. Has seen a dentist within 90 days prior to enrollment and been cleared to receive bone-strengthening agents.
6. Availability of a representative formalin fixed, paraffin embedded tumor specimen or fresh frozen tissue specimen that enables the definitive diagnosis of RCC, accompanied by an associated pathology report. If stored specimens are not available, an optional biopsy may be performed and specimens can be collected by surgical resection or biopsy of the primary tumor or biopsy or resection of a metastatic lesion.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
8. Demonstrates adequate organ function as defined below within 14 days prior to first study treatment:

   1. Absolute neutrophil count (ANC) >=1,500/ μL (without granulocyte colony stimulating factor support within 2 weeks prior to Cycle 1, Day 1).
   2. Platelets ≥100,000/ μL (without transfusion within 2 weeks prior to Cycle 1, Day 1).
   3. White Blood Cell count (WBC) counts ≥ 2500/μL.
   4. Lymphocyte count ≥ 500/μL.
   5. Hemoglobin ≥9.0 g/dL.

      Participants may be transfused or receive erythropoietic treatment to meet this criterion:
   6. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN). Participants with known Gilbert disease who have serum bilirubin level <= 3 x ULN may be enrolled.
   7. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) ≤2.5 X institutional upper limit of normal.
   8. Alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) ≤2.5 X institutional upper limit of normal.
   9. Alkaline phosphatase ≤2.5 X institutional upper limit of normal. For participants with documented liver metastases: AST and/or ALT ≤ 5 x ULN. For participants with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN.
   10. Creatinine ≤ 1.5 x within institutional upper limit of normal OR creatinine clearance ≥ 40 mL/min by institutional standard AND urine protein-creatinine ratio (UPCR) 1mg/mg.
   11. International Normalized Ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. This applies only to participants who are not receiving therapeutic anticoagulation; participants receiving therapeutic anticoagulation should be on a stable dose.
   12. Serum ionized calcium above lower limit of normal and ≤ 1.5 x ULN.
9. If any Grade ≥1 toxicities occurred in relation to prior treatment, patients must have recovered to baseline or ≤ Grade 1 unless adverse events are clinically insignificant or stable on supportive medication if needed.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
12. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
13. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
14. Sexually active fertile subjects and their partners must agree to use highly effective method of contraception (defined in Appendix 4) during the course of the study and for the following durations after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (e.g., condom), is required. In addition, men must agree not to donate sperm and women must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods.

    a. Through 186 days after the last dose of zanzalintinib for women of childbearing potential (WOCBP) or through 96 days after the last dose of zanzalintinib for men.
15. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria is met: permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone (FSH) level > 40 milli-international units per millilitre (mIU/mL) to confirm menopause). Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff. Exception: women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus).

Exclusion Criteria:

1. Prior treatment with zanzalintinib for RCC.
2. Receipt of any small molecule kinase inhibitor (including investigational) or vascular endothelial growth factor (VEGF)-targeted therapy within 2 weeks before the first dose of study treatment.
3. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
4. Participants requiring whole brain radiotherapy (WBRT).
5. Incomplete healing from prior radiotherapy as determined by the treating radiation oncologist or treating investigator.
6. Participation in an experimental drug study within 28 days of study enrollment.
7. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
8. Pregnant and lactating women are excluded from this study because zanzalintinib is an investigational product with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with zanzalintinib, breastfeeding should be discontinued if the mother is treated with zanzalintinib.
9. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1.
10. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation); Clinically significant hematuria, hematemesis, or hemoptysis of >0.5 tsp (2.5ml) of red blood or other history of significant bleeding within 12 weeks before first dose of study treatment.
11. Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
12. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
13. Concomitant anticoagulation with coumarin agents, direct thrombin inhibitors, factor Xa inhibitor betrixaban, or platelet inhibitors. Other anticoagulants are allowed.

    1. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    2. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.

    i. Participants who have known brain metastases and who require therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban are not eligible for this study.

    ii. Participants with known brain metastases and who are taking prophylactic low-dose aspirin for cardioprotection or low-dose (prophylactic-dose) low molecular weight heparin are eligible.

    Note: Subjects must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.
14. Previously identified allergy or hypersensitivity to components of the treatment.
15. Malignancy that requires anti-cancer directed therapy within the last 3 years. Exceptions include those cancers that are considered cured by local therapy (e.g. Basal cell carcinoma, squamous cell carcinoma, ductal carcinoma in situ of breast, bladder, or cervix) or other cancers that have low malignant potential and do not require systemic therapy (e.g. Gleason grade <6 prostate adenocarcinoma).
16. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
17. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
18. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of enrollment. Note: Base of skull lesions without definitive evidence of dural or brain parenchymal involvement are allowed.
19. Any complementary medications (e.g., herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
20. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    1. Congestive heart failure New York Heart Association Class 3 or 4, class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (e.g., ventricular flutter, ventricular fibrillation, Torsades de pointes).
    2. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    3. Stroke (including transient ischemic attack (TIA)), myocardial infarction, or other clinically significant arterial thrombotic and/or ischemic event within 6 months before first dose of study treatment.
    4. Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous events within 3 months before first dose of study treatment.

       Note: Subjects with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.

       Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.
    5. Prior history of myocarditis.
    6. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    i. Tumors invading the GI-tract from external viscera. ii. Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis.

    iii. Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months before first dose unless cause of obstruction is definitively managed and subject is asymptomatic.

    iv. Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.

    v. Known gastric or esophageal varices. vi. Ascites, pleural effusion, or pericardial fluid requiring drainage in last 4 weeks.
21. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 mL) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
22. Symptomatic cavitating pulmonary lesion(s) or endobronchial disease (asymptomatic or radiated lesions allowed).
23. Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta. Note: Subjects with intravascular tumor extension (e.g., tumor thrombus in renal vein or inferior V. cava) may be eligible following Principal Investigator approval.
24. Other clinically significant disorders that would preclude safe study participation.

    1. Active infection requiring systemic treatment. Note: Prophylactic antimicrobial treatments (antibiotics, antimycotic, antiviral) are allowed.
    2. Known infection with acute or chronic hepatitis B or C, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness except for subjects meeting all of the following criteria: (1) on stable anti-retroviral therapy; (2) Cluster of differentiation 4 positive (CD4+) T cell count ≥ 200/µL; and (3) an undetectable viral load. Note: HIV testing will be performed at screening if and as required by local regulation. Note: To be eligible, participants taking Cytochrome P450, family (CYP) inhibitors (e.g., zidovudine, ritonavir, cobicistat, didanosine) or Cytochrome P450, family 3 (CYP3) inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose. Note: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider.
    3. Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.

    i. Complete healing of intra-abdominal abscess must be confirmed before the first dose of study treatment d. Malabsorption syndrome. e. Pharmacologically uncompensated, symptomatic hypothyroidism. f. Moderate to severe hepatic impairment (Child-Pugh B or C). g. Requirement for hemodialysis or peritoneal dialysis. h. History of solid organ or allogeneic stem cell transplant.
25. Major surgery (as defined in Section 6.6.2.3; e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (i.e. nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (e.g., simple excision, tooth extraction) within 5 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment.

    Note: Fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
26. Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment.

    Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.
27. History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
28. Patients who are ineligible for CT contrast AND who are unable to undergo MRI for any reason.
29. Inability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube.
30. Other conditions, which in the opinion of the Investigator, would compromise the safety of the participant or the participant's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who have not progressed at 12 months (PFS12) | Up to 12 months
  The proportion of participants who have not demonstrated radiographic progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or demonstrated clinical progression-free survival (PFS) at 12 months after the start of study treatment. Twelve-month landmark PFS rate will be obtained with 95% confidence interval using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Percentage of participants with Skeletal Related Events (SRE) | Up to 24 months
  The percentage of participants who demonstrate an SREs defined as: 1) pathological fracture; 2) surgery or radiation to the bone; or 3) cord compression, by bone scan will be reported
Percentage of participants with osteonecrosis of the jaw (ONJ) | Up to 24 months
  The percentage of participants who demonstrate ONJ, by clinical exam will be reported.
Percentage of participants with reported treatment-related, systemic, adverse events | Up to 24 months
  The percentage of participants with treatment-related, systemic toxicity of any grade as classified by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported.
Median PFS | Up to 24 months
  PFS is defined as the time from day of study treatment initiation (C1D1) until evidence of disease progression per RECIST v1.1 criteria, in patients with measurable disease at baseline, or death from any cause. Participants will be censored for PFS at the start of any subsequent therapy or at last negative scan if there is no evidence of disease progression. The median PFS in months will be reported with a 95% confidence interval.
Median Overall Survival (OS) | Up to 24 months
  Overall survival (OS) will be defined starting from study treatment initiation (C1D1) until death from any cause or last follow-up. OS will be assessed using the Kaplan-Meier method and median OS in months will be reported with a 95% confidence interval.
Objective Response Rate (ORR) | Up to 24 months
  Objective response rate will be assessed in the measurable disease population only and is defined as the proportion of participants with either a demonstrated radiographic complete response ((CR); Disappearance of all target lesions and no new lesions)) or partial response ((PR); At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, and no appearance of new lesions)) according to RECIST v1.1 criteria. The proportion of all participants with 95% confidence interval will be reported.
Proportion of participants who have not progressed at 24 months (PFS24) | Up to 24 months
  The proportion of participants who have not demonstrated radiographic progression as defined by RECIST v1.1 or demonstrated clinical PFS at 24 months after the start of study treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Fitzgerald, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with study collaborators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: During the course of the study